CLINICAL TRIAL: NCT04064437
Title: Prevalence of Vertebral Fractures in Patients With Type 1 Diabetes (Diabetes Spine Fractures, DenSiFy)
Brief Title: Prevalence of Vertebral Fractures in Patients With Type 1 Diabetes
Acronym: DenSiFy
Status: Completed | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Claudia Gagnon, MD, CHU de Quebec-Universite Laval
Other Study IDs: 2019-4550
Record Dates: First submitted 2019-08-17; First posted 2019-08-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1; Bone Fracture; Bone Health
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Fractures, Bone | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with type 1 diabetes
  Interventions: Diagnostic Test: Clinical tests; Diagnostic Test: Biochemical tests; Diagnostic Test: DXA scan; Diagnostic Test: AGE Reader
- Healthy controls
  Interventions: Diagnostic Test: Clinical tests; Diagnostic Test: Biochemical tests; Diagnostic Test: DXA scan; Diagnostic Test: AGE Reader

INTERVENTIONS:
Diagnostic Test: Clinical tests — The investigators perform the following clinical tests: vibration threshold test, monofilament test, and height, weight and waist circumference measurement in every participant.
  Groups: Individuals with type 1 diabetes
Diagnostic Test: Clinical tests — The investigators perform the following clinical tests: height, weight and waist circumference measurement in every participant.
  Groups: Healthy controls
Diagnostic Test: Biochemical tests — The investigators perform blood and urine tests in every participant.
Diagnostic Test: DXA scan — The investigators perform a dual energy x-ray absorptiometry (DXA scan or osteodensitometry) in every participant.
Diagnostic Test: AGE Reader — The investigators perform a skin advanced glycation end products (AGEs) measurement with the AGE Reader machine in every participant.

SUMMARY:
Background : Type 1 diabetes is associated with an increased risk of fractures. The mechanisms accounting for this bone fragility are not yet fully understood. The lower bone mineral density (BMD) observed in individuals with type 1 diabetes cannot solely explain the higher fracture incidence. Bone microarchitecture defects significantly contribute to bone fragility. Few studies assessed spine fractures in type 1 diabetes.

This cross-sectional multicenter case-control study aims (1) to evaluate the prevalence of asymptomatic vertebral fractures in individuals with type 1 diabetes in comparison to age- and sex-matched healthy controls; (2) to compare individuals with diabetes with vertebral fractures and those without vertebral fracture using clinical, biochemical and radiological parameters.

ELIGIBILITY:
Individuals with type 1 diabetes

Inclusion Criteria:

* Diagnosis of type 1 diabetes for at least 5 years;
* Age 20 years and older.

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Conditions associated with bone disease (significant liver disease, intestinal malabsorption other than celiac disease, organ transplant, active cancer, rheumatoid arthritis, hyperthyroidism, hypothyroidism with abnormal thyroid-stimulating hormone (TSH), hyperparathyroidism, hypoparathyroidism, acromegaly, Cushing syndrome, adrenal insufficiency);
* Any of these medications in the past 6 months : glucocorticoids ≥ 7,5 mg prednisone/day or equivalency ≥ 3 months, aromatase inhibitors, antiandrogens, antiepileptic drugs, anticoagulants, sodium-glucose cotransporter-2 (SGLT-2) inhibitors, thiazolidinediones;
* Past medical history of traumatic vertebral fracture;
* Inability to consent.

Healthy controls

Inclusion Criteria:

* Age 20 years and older.

Exclusion Criteria:

* As above (as individuals with diabetes), and :
* Diagnosis of diabetes or prediabetes;
* Celiac disease;
* Chronic kidney disease (CrCl < 60 mL/min);
* Any of theses medications in the past 6 months : biphosphonates, teriparatide, denosumab, calcitonin;
* Past medical history of fragility fracture.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 127 individuals with type 1 diabetes and 64 healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Vertebral fracture detected with VFA | Baseline
  Vertebral Fracture Assessment (VFA) software of dual-energy X-ray absorptiometry (DXA scan) is used to identify vertebral fractures. If there is evidence of a vertebral fracture on VFA, a lateral and anteroposterior spine X-ray will be obtained to confirm the VFA results.

SECONDARY OUTCOMES:
Areal bone mineral density of the spine in g/cm2 | Baseline
  Measured by DXA scan
Areal bone mineral density of the spine, T-score | Baseline
  Measured by DXA scan
Areal bone mineral density of the spine, Z-score | Baseline
  Measured by DXA scan
Areal bone mineral density of proximal femur in g/cm2 | Baseline
  Measured by DXA scan
Areal bone mineral density of proximal femur, T-score | Baseline
  Measured by DXA scan
Areal bone mineral density of proximal femur, Z-score | Baseline
  Measured by DXA scan
Areal bone mineral density of total hip in g/cm2 | Baseline
  Measured by DXA scan
Areal bone mineral density of total hip, T-score | Baseline
  Measured by DXA scan
Areal bone mineral density of total hip, Z-score | Baseline
  Measured by DXA scan
Areal bone mineral density of distal radius in g/cm2 | Baseline
  Measured by DXA scan
Areal bone mineral density of distal radius, T-score | Baseline
  Measured by DXA scan
Areal bone mineral density of distal radius, Z-score | Baseline
  Measured by DXA scan
Lean mass (arm, leg, trunk, android, gynoid and total) | Baseline
  Body composition measured by DXA scan
Fat mass (arm, leg, trunk, android, gynoid and total) | Baseline
  Body composition measured by DXA scan
Skin AGE measurement | Baseline
  Measured by AGE Reader
C-telopeptide | Baseline
  Bone turnover marker (serum)
Sclerostin | Baseline
  Bone turnover marker (serum)
Osteocalcin | Baseline
  Bone turnover marker (serum)

OTHER OUTCOMES:
HbA1C | Baseline
  Diabetes control marker
Hemoglobin | Baseline
  Blood level measurement
Creatinine | Baseline
  Blood level measurement
Lipid panel | Baseline
  Blood level measurement
Thyroid-stimulating hormone (TSH) | Baseline
  Blood level measurement
Calcium | Baseline
  Blood level measurement
Albumine | Baseline
  Blood level measurement
Phosphate | Baseline
  Blood level measurement
25-Hydroxyvitamin D | Baseline
  Blood level measurement
Parathormone (PTH) | Baseline
  Blood level measurement
Insulin like growth factor-1 (IGF-1) | Baseline
  Blood level measurement
Antitransglutaminase antibodies | Baseline
  Blood level measurement
Immunoglobulin A (IgA) | Baseline
  Blood level measurement
Follicle stimulating hormone (FSH, women) | Baseline
  Blood level measurement
Total testosterone (men) | Baseline
  Blood level measurement
Sex hormone-binding globulin (SHBG, men) | Baseline
  Blood level measurement
Microalbuminuria | Baseline
  Urine microalbuminuria / urine creatinine ratio measurement

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, Dr, Principal Investigator — CHU de Québec - Université Laval
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal (IRCM), Montreal, Quebec
  - Centre de recherche du CHU de Québec - Université Laval, Québec

REFERENCES:
- [Result] Coll JC, Garceau E, Leslie WD, Genest M, Michou L, Weisnagel SJ, Mac-Way F, Albert C, Morin SN, Rabasa-Lhoret R, Gagnon C. Prevalence of Vertebral Fractures in Adults With Type 1 Diabetes: DenSiFy Study (Diabetes Spine Fractures). J Clin Endocrinol Metab. 2022 Apr 19;107(5):e1860-e1870. doi: 10.1210/clinem/dgac031. PMID 35090169